CLINICAL TRIAL: NCT04924283
Title: Effects of a Cognitive Interference Task on Alcohol Craving and Consumption Among Women
Brief Title: Cognitive Interference Task on Alcohol Craving and Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christine Hahn, Research Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00102351
Record Dates: First submitted 2021-06-06; First posted 2021-06-11 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Drinking; Craving
Keywords: ecological momentary assessment; cognitive interference
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Interference Task (Experimental): Participants in this arm will complete random assessments of alcohol use and cravings on their phone, and be prompted to play Tetris on their phone after reporting cravings for alcohol.
  Interventions: Behavioral: Tetris and Assessments
- Assessment Only (Active Comparator): Participants in this arm will complete random assessments of alcohol use and cravings on their phone.
  Interventions: Other: Assessment Only

INTERVENTIONS:
Behavioral: Tetris and Assessments — Participants will complete assessments on their phone to rate cravings for alcohol. Participants will complete a visual cognitive interference task (i.e., play Tetris on their phone) after endorsing a alcohol craving, and then re-rate craving after the task.
  Arms: Cognitive Interference Task
Other: Assessment Only — Participants will complete assessments on their phone to rate cravings for alcohol.
  Arms: Assessment Only

SUMMARY:
The purpose of this study is to test a brief task of playing the game Tetris to reduce alcohol cravings and alcohol use. Women who are seen at primary care and recruited through the community will be asked to rate alcohol craving and use for a 1-week baseline period. Then they will be randomly assigned to play the Tetris game on their phones daily or to a control condition for a 2-week period. Participants will also complete a cue-reactivity task, that involves viewing pictures of alcohol and rating cravings.

ELIGIBILITY:
Inclusion Criteria:

1. Female, any race or ethnicity, age 21 to 65 years old.
2. Able to comprehend English.
3. At least one heavy drinking per week (i.e., consuming at least four or more drinks in one day) for the last two weeks
4. Internet access and reliable electronic device

Exclusion Criteria:

1. More than four heavy drinking days per week.
2. Currently engaged in treatment for Alcohol Use Disorder (AUD).
3. Current clinically significant bipolar affective disorder, schizophrenia, or psychotic disorder.
4. Pregnant.
5. Imminently suicidal or homicidal.
6. Participants taking psychoactive medications that may affect alcohol craving or consumption.
7. A score of 10 or higher on the Clinical Institute of Alcohol Withdrawal Revised (CIWA-R).24

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female-ADD RATIONALE
Enrollment: 40 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Interference Task: Participants in this arm will complete random assessments of alcohol use and cravings on their phone, and be prompted to play Tetris on their phone after reporting cravings for alcohol.
  Tetris and Assessments: Participants will complete assessments on their phone to rate cravings for alcohol. Participants will complete a visual cognitive interference task (i.e., play Tetris on their phone) after endorsing a alcohol craving, and then re-rerate craving after the task.
Period: Overall Study
Arm/Group | Cognitive Interference Task | Assessment Only
Started | 20 | 20
Completed | 20 | 17
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Interference Task | Assessment Only | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.90 (9.67) | 29.90 (7.80) | 30.40 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 17 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Craving
Description: Participants completed the 4-item imagery subscale of the Craving Experiences Questionnaire, which measures craving/intense desire. Items are rated on a 0 to 10 point scale. A mean was calculated from the 4-item imagery subscale, with a possible range of 0 to 10. Higher scores indicate greater alcohol craving.
Time Frame: Participants reported cravings one-month after the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
units on a scale | 2.51 (2.65) | 2.79 (2.57)

2. Primary Outcome: Average Drinks Per Occasion
Description: Participants completed the Timeline Follow Back, which assesses past-month alcohol consumption. The outcome measure is average drinks per drinking occasion. Scores ranged from 0 to 6.29 drinks. Higher scores indicate greater average drinks consumed per occasion.
Time Frame: Participants reported alcohol consumption one month after the intervention.
Measure: Mean (Standard Deviation); unit: average drinks per drinking occasion
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
average drinks per drinking occasion | 3.31 (1.62) | 2.75 (1.38)

3. Primary Outcome: Number of Standard Drinks
Description: Participants reported the number of standard drinks consumed yesterday. The scale ranged from 0 to more than 20. Higher scores indicate more drinks consumed. A single value for number of standard drinks reported each day for 14 days was averaged across all participants.
Time Frame: Participants reported number of standard drinks each morning at a scheduled time for 14 days.
Measure: Mean (Standard Deviation); unit: drinks
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
drinks | 2.00 (2.87) | 1.58 (2.06)

4. Primary Outcome: Changes in Alcohol Craving Before and After Tetris Task
Description: During the intervention phase, participants received up to three daily random in-vivo assessments assessing craving. Participants in the experimental group completed a Tetris task if they reported a positive response to craving and participants in the control group took an equivalently long break. Participants then re-rated their craving. Both craving assessments used a single item from the Visual Analogue Craving Scale ("How strong is your craving for alcohol RIGHT NOW?"), ranging from 0 to 100. The outcome measure represents change in craving, calculated as post-task craving minus pre-task craving. The change score was the difference in craving before and after the experimental task or the wait period. A single value for change in alcohol craving reported at each assessment during the 14 days was averaged across all participants.
Time Frame: Participants reported pre- and post-task alcohol craving up to three times per day for a 14-day intervention period. Post-task craving was measured right after the Tetris task/control break and pre-task craving was measured directly before.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
units on a scale | -10.16 (20.56) | -2.63 (13.95)

5. Primary Outcome: Changes in Alcohol Craving Before and After Cue Tetris Task
Description: During the intervention phase, participants received a daily Cue Reactivity Ecological Momentary Assessment (CREMA), which provides real-time responses to alcohol-related imagery. After the CREMA, participants in the experimental group completed a Tetris task and participants in the control group took an equivalently long break. Participants then re-rated their craving. Both craving assessments used a single item from the Visual Analogue Craving Scale ("How strong is your craving for alcohol RIGHT NOW?"), ranging from 0 to 100. The outcome measure represents change in craving, calculated as post-task craving minus pre-task craving. A single value for change in alcohol craving reported at each cue reactivity assessment during the 14 days was averaged across all participants.
Time Frame: Participants reported pre- and post-task alcohol craving up to once a day for a 14-day intervention period. Post-task craving was measured right after the CREMA/wait period and pre-task craving was measured directly before.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
units on a scale | 0.30 (17.93) | 1.69 (12.47)

6. Secondary Outcome: Obsessive Thoughts About Alcohol
Description: Participants rated their craving and drinking behavior on the 6-item Obsessive subscale of the Obsessive Compulsive Drinking Scale, which measures obsessive thoughts about alcohol. Each item is provided on a scale from 0 to 4. A total score was calculated, with a range of 0 to 24. Higher scores represent more obsessive thoughts of drinking.
Time Frame: Participants reported obsessive thoughts about alcohol at a single baseline assessment, which occurred the day before the EMA period began.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
units on a scale | 4.10 (3.77) | 2.55 (2.44)

7. Secondary Outcome: Drinking Motives
Description: Participants rated their motivations for drinking alcohol on the Drinking Motives Questionnaire. The Drinking Motives Questionnaire consists of 28 items, each rated on a 1 to 5 scale. A mean score was calculated using all 28 items, with a total score range of 1 to 5. Higher scores indicate higher endorsement of motives to drink alcohol.
Time Frame: Participants reported drinking motives at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
score on a scale | 2.251786 (.6690041) | 2.198214 (.6381906)

8. Secondary Outcome: Feasibility of Intervention
Description: The percentage of prompts participants responded to, calculated by the number of surveys participants responded to divided by the number of all possible surveys multiplied by 100%. Higher numbers indicate a greater number of responses.
Time Frame: This was recorded during the 14-day intervention phase.
Population: Surveys during the 14-day intervention phase. Each participant was sent 4 surveys per day for 14 days.
Measure: Number; unit: percentage of possible surveys completed
Units Other Than Participants: surveys
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
Number analyzed (surveys) | 1120 | 1120
percentage of possible surveys completed | 89.4 | 86.3

9. Secondary Outcome: Acceptability Ratings
Description: Participants rated acceptability of the intervention on the Acceptability of Intervention Measure. Each item was rated on a 1 to 5 point scale. Total scores of 4 items were calculated with higher scores indicating greater acceptability (range 4-20).
Time Frame: Recorded within one-week after the intervention.
Population: Only the experimental group rated acceptability of playing Tetris because the control did not play the game.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 0
units on a scale | 14.3 (4.243881) |

10. Other Pre Specified Outcome: Mood Ratings
Description: Participants will rate their mood on a 100-point scale ranging from unpleasant to pleasant. A higher score indicates a better or more pleasant mood.
Time Frame: This will be recorded during the intervention phase.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Stress Ratings
Description: Participants will rate their stress using a 100-point scale ranging from not at all to extremely. A higher score indicates greater stress.
Time Frame: This will be recorded during the intervention phase.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Depression Symptoms
Description: Participants responded to the Patient Health Questionnaire assessing symptoms of depression. The item assessing suicidal ideation was omitted. The 8 items included were rated on a 4 point scale ranging from 0 to 3 and totaled. Scores ranged from 0 to 24 and higher scores indicate greater symptoms of depression.
Time Frame: Participants reported depression symptoms at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
score on a scale | 5.25 (3.971941) | 5.75 (5.087394)

13. Other Pre Specified Outcome: Post-traumatic Stress Disorder Symptoms
Description: Participants rated symptoms of posttraumatic stress disorder on the Posttraumatic Stress Disorder Checklist for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5). Each symptom is rated on a 0 to 4 point scale. The 20 items are totaled and scores can range from 0 to 80. Higher scores indicate greater posttraumatic stress disorder symptoms.
Time Frame: Participants reported posttraumatic stress symptoms at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
score on a scale | 17.9 (14.06) | 15.85 (14.92)

14. Other Pre Specified Outcome: Alcohol Use Disorder Symptoms at Baseline
Description: Participants rated symptoms of alcohol use disorder on the the Alcohol Use Disorder Identification Test (AUDIT). The AUDIT includes ten items assessing symptoms of alcohol use disorder. Each item is rated from 0 to 4 and items are added. Total scores on the Alcohol Use Disorder Identification Test (AUDIT) are reported. A score of 8 or higher is the suggested cut-off for harmful drinking.
Time Frame: Participants reported self-reported symptoms of alcohol use disorder at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
score on a scale | 12.3 (6.681475) | 10.4 (7.214021)

15. Other Pre Specified Outcome: Alcohol Use Disorder at Baseline
Description: Participants completed a structured interview to assess alcohol use disorder symptoms using the DIAMOND. The percent of participants who met criteria for an alcohol use disorder based on a clinical interview is reported.
Time Frame: Participants reported alcohol use disorder symptoms at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
Participants | 12 | 11

16. Other Pre Specified Outcome: COVID-19 Related Stress at Baseline
Description: Participants reported the impact of coronavirus disease 2019 (COVID-19) on stress and drinking. Average of self-reported stress due to COVID-19 on a single item rated on a 4 point scale (0 to 4) is reported. Higher scores indicate greater stress.
Time Frame: Participants reported COVID-19 related stress at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
units on a scale | 1.65 (1.089423) | 1.5 (1.147079)

17. Other Pre Specified Outcome: Impulsivity at Baseline
Description: Participants reported impulsivity on the Short Negative Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency Impulsive Behavior Scale. The total scores for negative urgency is reported. Total scores were calculated for negative urgency (range 4 to 16) by adding 4 items assessing tendency to act rashly when feeling upset. Each item was rated on a 1 to 4 scale, with higher scores indicating greater tendency to act rashly when upset.
Time Frame: Participants reported impulsivity at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Interference Task | Assessment Only
Number analyzed (Participants) | 20 | 20
score on a scale | 11.5 (2.800376) | 11.7 (3.599708)

ADVERSE EVENTS:
Time Frame: Potential adverse events were collected during a 15 month period.
Description: It does not differ.
Arm/Group | Cognitive Interference Task | Assessment Only
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04924283/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT04924283/ICF_002.pdf